CLINICAL TRIAL: NCT02528214
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dupilumab in Patients With Severe Steroid Dependent Asthma
Brief Title: Evaluation of Dupilumab in Patients With Severe Steroid Dependent Asthma
Acronym: VENTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC13691; 2015-001573-40 (EudraCT Number); U1111-1170-7152 (Other: UTN)
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2017-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Prednisone; Prednisolone; Therapeutics; Albuterol; Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo q2w (Placebo Comparator): 2 subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1, followed by a single injection every 2 weeks (q2w) for 24 weeks in combination with OCS - (prednisone or prednisolone) and stable inhaled corticosteroid (ICS). OCS dose was reduced according to a predetermined titration schedule every 4 weeks until Week 20. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
  Interventions: Drug: Placebo; Drug: Oral corticosteroid therapy (prednisone/prednisolone); Drug: Inhaled corticosteroid (ICS) therapy; Drug: Albuterol/Salbutamol; Drug: Levalbuterol/Levosalbutamol
- Dupilumab 300 mg q2w (Experimental): 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection q2w for 24 weeks in combination with OCS - (prednisone or prednisolone) and stable ICS. OCS dose was reduced according to a predetermined titration schedule every 4 weeks until Week 20. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: Oral corticosteroid therapy (prednisone/prednisolone); Drug: Inhaled corticosteroid (ICS) therapy; Drug: Albuterol/Salbutamol; Drug: Levalbuterol/Levosalbutamol

INTERVENTIONS:
Drug: Dupilumab — Solution for injection, Subcutaneous injection in the abdomen, upper thigh or upper arm.
  Other Names: REGN668; SAR231893
  Arms: Dupilumab 300 mg q2w
Drug: Placebo — Solution for injection, Subcutaneous injection in the abdomen, upper thigh or upper arm.
  Arms: Placebo q2w
Drug: Oral corticosteroid therapy (prednisone/prednisolone) — Oral administration.
Drug: Inhaled corticosteroid (ICS) therapy — Oral inhalation, stable dose (high dose) of ICS in combination with up to 2 other controller medicines (second or third controller therapy).
Drug: Albuterol/Salbutamol — Oral inhalation as needed.
Drug: Levalbuterol/Levosalbutamol — Oral inhalation as needed.

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab, compared with placebo, for reducing the use of maintenance oral corticosteroids (OCS) in participants with severe steroid-dependent asthma.

Secondary Objectives:

* To evaluate the safety and tolerability of dupilumab.
* To evaluate the effect of dupilumab in improving participants-reported outcomes.
* To evaluate dupilumab systemic exposure and the incidence of treatment-emergent antidrug antibodies.

DETAILED DESCRIPTION:
The total study duration per participant was up to 46 weeks, consisting of a screening period of 3 to up to 8 weeks (up to 10 weeks for participants who experienced a clinically significant asthma exacerbation during the screening period), a randomized treatment period of up to 24 weeks, and a post-treatment period of 12 weeks.

Participants who completed treatment were considered for eligibility into the long term extension study LTS12551 (NCT02134028).

ELIGIBILITY:
Inclusion criteria :

Adult and adolescent (12 years of age or older) participants with a physician diagnosis of asthma for >=12 months, based on the Global Initiative for Asthma (GINA) 2014 guidelines and the following criteria:

* Participants with severe asthma and a well-documented, regular prescribed treatment of maintenance corticosteroids in the 6 months prior to Visit 1 and using a stable OCS dose (ie, no change of OCS dose) for 4 weeks prior to Visit 1. Participants must be taking 5 to 35 mg/day of prednisone/prednisolone, or the equivalent, at Visit 1 and at the randomization visit. In addition, the participants must agree to switch to study-required prednisone/prednisolone as their OCS and use it per protocol for the duration of the study.
* Existing treatment with high-dose inhaled corticosteroid (ICS; >500 mcg total daily dose of fluticasone propionate or equivalent) in combination with a second controller (ie, long-acting beta agonist [LABA], leukotriene receptor antagonist [LTRA]) for at least 3 months with a stable dose of ICS for >=1 month prior to Visit 1. In addition, participants requiring a third controller for their asthma are considered eligible for this study, and it should also be used for at least 3 months with a stable dose >= 1 month prior to Visit 1.
* A forced expiratory volume in 1 second (FEV1) <80% of predicted normal for adults and <=90% of predicted normal for adolescents at Visit 1.
* Evidence of asthma as documented by either: reversibility of at least 12% and 200 mL in FEV1 after the administration of 200 to 400 mcg (2 to 4 inhalations of albuterol/salbutamol or levalbuterol/levosalbutamol, or of a nebulized solution of albuterol/salbutamol or levalbuterol/levosalbutamol, if considered as a standard office practice) before randomization or documented in the 12 months prior to Visit 1 OR airway hyperresponsiveness (methacholine: provocative concentration that causes a positive reaction [PC20] of <8 mg/mL) documented in the 12 months prior to Visit 1.

Exclusion criteria:

* Participants <12 years of age or the minimum legal age for adolescents in the country of the investigative site, whichever is higher (for those countries where local regulations permit enrollment of adults only, participant recruitment will be restricted to those who were >=18 years of age).
* Participants who weighed <30.0 kg.
* Chronic obstructive pulmonary disease (COPD) or other lung diseases (eg, idiopathic pulmonary fibrosis, Churg-Strauss Syndrome, allergic bronchopulmonary aspergillosis, cystic fibrosis) which may impair lung function.
* Clinical evidence or imaging (eg, chest X-ray, computed tomography, magnetic resonance imaging) within 12 months of Visit 1 with clinically significant findings of lung disease(s) other than asthma, as per local standard of care.
* A participant who experiences a deterioration of asthma that results in emergency treatment or hospitalization within 4 weeks of Screening Visit 1.
* A participant who requires 12 puffs or more of rescue medication on any 1 day in the week prior to Visit 1.
* A participant who has experienced an upper or lower respiratory tract infection within the 4 weeks prior to screening.
* Current smoker or cessation of smoking within 6 months prior to Visit 1.
* Previous smoker with a smoking history >10 pack-years.
* Comorbid disease that might interfere with the evaluation of the investigational medicinal product.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-10-15; Primary Completion 2017-09-20 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (80):
- United States (8):
  - Investigational Site Number 840022, Los Angeles, California
  - Investigational Site Number 840014, Rolling Hills Estates, California
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840010, Pittsburgh, Pennsylvania
  - Investigational Site Number 840062, Amarillo, Texas
  - Investigational Site Number 840070, McKinney, Texas
  - Investigational Site Number 840128, McKinney, Texas
  - Investigational Site Number 840118, Plano, Texas
- Argentina (3):
  - Investigational Site Number 032003, Buenos Aires
  - Investigational Site Number 032001, Caba
  - Investigational Site Number 032091, Caba
- Belgium (3):
  - Investigational Site Number 056002, Brussels
  - Investigational Site Number 056003, Ghent
  - Investigational Site Number 056001, Leuven
- Brazil (3):
  - Investigational Site Number 076013, São Bernardo do Campo
  - Investigational Site Number 076011, São Paulo
  - Investigational Site Number 076002, Sorocaba
- Canada (6):
  - Investigational Site Number 124009, Calgary
  - Investigational Site Number 124016, Hamilton
  - Investigational Site Number 124003, Mississauga
  - Investigational Site Number 124013, Ottawa
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124017, Vancouver
- Chile (3):
  - Investigational Site Number 152007, Quillota
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152008, Talca
- Colombia (2):
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170006, Bogotá
- Hungary (2):
  - Investigational Site Number 348301, Balassagyarmat
  - Investigational Site Number 348303, Edelény
- Israel (5):
  - Investigational Site Number 376003, Haifa
  - Investigational Site Number 376001, Kfar Saba
  - Investigational Site Number 376005, Petah Tikva
  - Investigational Site Number 376002, Rehovot
  - Investigational Site Number 376004, Tel Litwinsky
- Italy (6):
  - Investigational Site Number 380005, Catania
  - Investigational Site Number 380002, Genova
  - Investigational Site Number 380008, Napoli
  - Investigational Site Number 380009, Palermo
  - Investigational Site Number 380001, Pisa
  - Investigational Site Number 380003, Reggio Emilia
- Mexico (5):
  - Investigational Site Number 484016, Acapulco
  - Investigational Site Number 484013, Chihuahua City
  - Investigational Site Number 484001, Guadalajara
  - Investigational Site Number 484002, Mexico City
  - Investigational Site Number 484003, Monterrey
- Netherlands (2):
  - Investigational Site Number 528001, Arnhem
  - Investigational Site Number 528002, Dordrecht
- Poland (5):
  - Investigational Site Number 616006, Bialystok
  - Investigational Site Number 616097, Krakow
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616010, Warsaw
  - Investigational Site Number 616011, Żnin
- Romania (7):
  - Investigational Site Number 642104, Bucharest
  - Investigational Site Number 642103, Bucharest
  - Investigational Site Number 642102, Cluj-Napoca
  - Investigational Site Number 642107, Cluj-Napoca
  - Investigational Site Number 642108, Cluj-Napoca
  - Investigational Site Number 642105, Timișoara
  - Investigational Site Number 642106, Timișoara
- Russia (5):
  - Investigational Site Number 643006, Moscow
  - Investigational Site Number 643007, Moscow
  - Investigational Site Number 643099, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643009, Saint Petersburg
- Spain (6):
  - Investigational Site Number 724014, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724013, Madrid
  - Investigational Site Number 724006, Pozuelo de Alarcón
  - Investigational Site Number 724007, Sant Boi de Llobregat
  - Investigational Site Number 724096, Santiago de Compostela
- Ukraine (9):
  - Investigational Site Number 804007, Chernivtsi
  - Investigational Site Number 804004, Ivano-Frankivsk
  - Investigational Site Number 804009, Ivano-Frankivsk
  - Investigational Site Number 804001, Kharkiv
  - Investigational Site Number 804003, Kyiv
  - Investigational Site Number 804011, Kyiv
  - Investigational Site Number 804006, Odesa
  - Investigational Site Number 804002, Poltava
  - Investigational Site Number 804019, Vinnytsia

REFERENCES:
- [Result] Rabe KF, Nair P, Brusselle G, Maspero JF, Castro M, Sher L, Zhu H, Hamilton JD, Swanson BN, Khan A, Chao J, Staudinger H, Pirozzi G, Antoni C, Amin N, Ruddy M, Akinlade B, Graham NMH, Stahl N, Yancopoulos GD, Teper A. Efficacy and Safety of Dupilumab in Glucocorticoid-Dependent Severe Asthma. N Engl J Med. 2018 Jun 28;378(26):2475-2485. doi: 10.1056/NEJMoa1804093. Epub 2018 May 21. PMID 29782224
- [Derived] Sher LD, Passalacqua G, Taille C, Cohn L, Daizadeh N, Pandit-Abid N, Soler X, Khodzhayev A, Jacob-Nara JA, Deniz Y, Rowe PJ, Nag A, Zhang Y. The long-term effect of dupilumab on dyspnea, sleep, and activity in oral corticosteroid-dependent severe asthma. Ann Allergy Asthma Immunol. 2023 Mar;130(3):298-304. doi: 10.1016/j.anai.2022.12.002. Epub 2022 Dec 9. PMID 36509407
- [Derived] Berger P, Menzies-Gow A, Peters AT, Kuna P, Rabe KF, Altincatal A, Soler X, Pandit-Abid N, Siddiqui S, Jacob-Nara JA, Deniz Y, Rowe PJ. Long-term efficacy of dupilumab in asthma with or without chronic rhinosinusitis and nasal polyps. Ann Allergy Asthma Immunol. 2023 Feb;130(2):215-224. doi: 10.1016/j.anai.2022.11.006. Epub 2022 Nov 7. PMID 36356712
- [Derived] Lugogo N, Mohan A. Are We Poised to Change the Trajectory of Maintenance Oral Corticosteroid Use in Severe Asthma in the Age of Biologics? Chest. 2022 Jul;162(1):4-5. doi: 10.1016/j.chest.2022.04.004. No abstract available. PMID 35809937
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Domingo C, Maspero JF, Castro M, Hanania NA, Ford LB, Halpin DMG, Jackson DJ, Daizadeh N, Djandji M, Mitchell CP, Crikelair N, Jacob-Nara JA, Deniz Y, Rowe PJ, Ortiz B. Dupilumab Efficacy in Steroid-Dependent Severe Asthma by Baseline Oral Corticosteroid Dose. J Allergy Clin Immunol Pract. 2022 Jul;10(7):1835-1843. doi: 10.1016/j.jaip.2022.03.020. Epub 2022 Apr 8. PMID 35398549
- [Derived] Sher LD, Wechsler ME, Rabe KF, Maspero JF, Daizadeh N, Mao X, Ortiz B, Mannent LP, Laws E, Ruddy M, Pandit-Abid N, Jacob-Nara JA, Gall R, Rowe PJ, Deniz Y, Lederer DJ, Hardin M. Dupilumab Reduces Oral Corticosteroid Use in Patients With Corticosteroid-Dependent Severe Asthma: An Analysis of the Phase 3, Open-Label Extension TRAVERSE Trial. Chest. 2022 Jul;162(1):46-55. doi: 10.1016/j.chest.2022.01.071. Epub 2022 Feb 22. PMID 35217003
- [Derived] Tohda Y, Matsumoto H, Miyata M, Taguchi Y, Ueyama M, Joulain F, Arakawa I. Cost-effectiveness analysis of dupilumab among patients with oral corticosteroid-dependent uncontrolled severe asthma in Japan. J Asthma. 2022 Nov;59(11):2162-2173. doi: 10.1080/02770903.2021.1996596. Epub 2021 Dec 8. PMID 34752208
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=29782224&report=abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 68 centers in 17 countries. A total of 390 participants were screened between October 2015 & April 2017, of which,210 were randomized & treated. 180 participants were screen failures mainly due to exclusion criteria met & inclusion criteria not met. Assignment was done by Interactive Voice/Web Response System(IVRS/IWRS).
Pre-assignment Details: Screening period included an OCS optimization phase (up to 10 weeks) where participants using OCS other than prednisone/prednisolone switched to these OCS. At the end of period, participants were randomized in 1:1 ratio (dupilumab:placebo).Randomization was stratified by optimized OCS dose (=<10 & >10 mg/day) at randomization visit & by country.
Groups:
- Placebo q2w: 2 subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1, followed by a single injection every 2 weeks (q2w) for 24 weeks in combination with OCS - (prednisone or prednisolone) and stable ICS. OCS dose was reduced according to a predetermined titration schedule every 4 weeks until Week 20.
- Dupilumab 300 mg q2w: 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection q2w for 24 weeks in combination with OCS - (prednisone or prednisolone) and stable ICS. OCS dose was reduced according to a predetermined titration schedule every 4 weeks until Week 20.
Period: Overall Study
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Started | 107 | 103
Treated | 107 | 103
Completed | 107 | 100
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Other than specified above | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Placebo q2w: 2 subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1, followed by a single injection q2w for 24 weeks in combination with OCS - (prednisone or prednisolone) and stable ICS. OCS dose was reduced according to a predetermined titration schedule every 4 weeks until Week 20.
- Total: Total of all reporting groups
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w | Total
Number analyzed (Participants) | 107 | 103 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.8) | 51.9 (12.5) | 51.3 (12.6)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 2 | 1 | 3
  Between 18 and 64 years | 88 | 91 | 179
  >=65 years | 17 | 11 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 62 | 127
  Male | 42 | 41 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 45
  Not Hispanic or Latino | 85 | 80 | 165
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 100 | 97 | 197
  Black/of African descent | 1 | 4 | 5
  Asian/Oriental | 2 | 0 | 2
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 2 | 1 | 3
Baseline Blood Eosinophil Count [Count of Participants; unit: Participants]
  <0.15 Giga/L | 38 | 22 | 60
  >=0.15 - <0.3 Giga/L | 28 | 33 | 61
  >=0.3 Giga/L | 41 | 48 | 89
Baseline Optimized Daily OCS Dose [Mean (Standard Deviation); unit: mg/day] — During screening period and before randomization, OCS dose was adjusted in each participant to achieve the lowest OCS dose, also known as optimized dose, required for management of participant's asthma.Participants using OCS medications other than prednisone/prednisolone were switched to either of these corticosteroids at a dose clinically comparable to their current stable OCS dose. To optimize the OCS dose, investigators were instructed to adjust the OCS dose weekly according to a pre-specified titration schedule, based on changes in participant's asthma control, and their clinical judgment.
  mg/day | 11.75 (6.31) | 10.75 (5.9) | 11.26 (6.12)
Daily OCS Dose at Visit 1 (i.e. preoptimization) [Mean (Standard Deviation); unit: mg/day] | 11.83 (6.02) | 11.79 (6.4) | 11.81 (6.20)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Reduction From Baseline in Oral Corticosteroids (OCS) Dose at Week 24 While Maintaining Asthma Control
Description: Percentage reduction of OCS dose was calculated as (optimized OCS dose [mg/day] at baseline - final OCS dose at Week 24)/optimized OCS dose at baseline x 100. Result is presented as Least Squares Mean (Standard Error) percentage reduction from baseline derived from ANCOVA model with missing data multiply imputed.
Time Frame: Baseline, Week 24
Population: Analysis was performed on intent-to-treat (ITT) population which included randomized population analysed according to the treatment group allocated by randomization regardless of whether the treatment kit was used or not.
Measure: Least Squares Mean (Standard Error); unit: Percentage reduction from baseline
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
Percentage reduction from baseline | 41.85 (4.57) | 70.09 (4.90)
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; The outcome measure was analyzed using analysis of covariance (ANCOVA) model which included percentage reduction of OCS dose at Week 24 as the response variable, and treatment group, baseline eosinophil level, optimized OCS dose at baseline, region as covariates. Missing data was imputed using a pattern mixture model by multiple imputation approach; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measure are reported and continued when previous outcome measure was statistically significant at two-sided 0.05. Only the primary and the first 4 secondary outcome measures were included in the procedure; p < 0.0001, ANCOVA — Threshold for significance at two-sided 0.05 level; Least Square (LS) Mean Difference = 28.24, 95% CI 2-sided [15.81 to 40.67] — LS mean difference represents reduction difference i.e. dupilumab - placebo

2. Primary Outcome: Supplementary Presentation of Primary Outcome Measure Data: Median Percentage Reduction From Baseline in Oral Corticosteroids Dose at Week 24 While Maintaining Asthma Control
Description: The Primary Outcome Measure (Percentage Reduction From Baseline in Oral Corticosteroids Dose at Week 24 While Maintaining Asthma Control) is summarized above, as LS Mean (SE). Table below provides a supplementary presentation of the Primary Outcome Measure data; result is presented as median (inter-quartile range). Percentage reduction of OCS dose was calculated as (optimized OCS dose [mg/day] at baseline - final OCS dose at Week 24)/optimized OCS dose at baseline x 100.
Time Frame: Baseline, Week 24
Population: Analysis population included ITT patients with available data.
Measure: Median (Inter-Quartile Range); unit: percentage reduction from baseline
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 106 | 101
percentage reduction from baseline | 50.0 [0 to 100.0] | 100.0 [62.5 to 100.0]

3. Secondary Outcome: Percentage of Participants Achieving >= 50% Reduction in Oral Corticosteroids Dose at Week 24 While Maintaining Asthma Control
Description: Participants were classified according to the binary status of whether or not the 50% OCS dose reduction criterion was achieved at week 24.
Time Frame: Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
percentage of participants | 53.3 | 79.6
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; The outcome measure was analyzed using a logistic regression model. The model included the binary status of whether or not a participant achieved the 50% OCS dose reduction criterion as the response variable, and treatment groups, optimized OCS dose at baseline, regions, and baseline eosinophil level subgroups as covariates. Missing data was imputed by using a pattern mixture model by multiple imputation approach; Test type: Superiority — Testing was performed according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant); p < 0.0001, Regression, Logistic — Threshold for significance at 0.05; Odds Ratio (OR) = 3.98, 95% CI 2-sided [2.06 to 7.67] — Dupilumab 300 mg q2w v Placebo q2w

4. Secondary Outcome: Percentage of Participants Achieving a Reduction in Oral Corticosteroids Dose to <5 mg/Day at Week 24 While Maintaining Asthma Control
Description: Participants were classified according to the binary status of whether or not the reduction of OCS dose to <5 mg/day was achieved at Week 24.
Time Frame: Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
percentage of participants | 37.4 | 71.8
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; The outcome measure was analyzed using a logistic regression model. The model included the binary status of whether or not a participant achieved a reduction of OCS dose to <5 mg/day at Week 24 as the response variable, treatment groups, optimized OCS dose at baseline, regions, and baseline eosinophil level subgroups as covariates. Missing data was imputed by using a pattern mixture model by multiple imputation approach; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05; Odds Ratio (OR) = 4.48, 95% CI 2-sided [2.39 to 8.39] — Dupilumab 300 mg q2w v Placebo q2w

5. Secondary Outcome: Percentage of Participants Achieving Maximum Possible Reduction in Oral Corticosteroids Dose Per Protocol at Week 24 While Maintaining Asthma Control
Description: For all participants except those with baseline OCS dose at 35 mg/day, the maximum possible reduction corresponds to reduction to 0 mg/day (no longer requiring OCS). For participants starting with 35 mg/day at baseline, the maximum possible reduction is 32.5 mg/day (i.e. minimum dose per protocol is 2.5 mg).
Time Frame: Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
percentage of participants | 29.9 | 52.4
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; The outcome was analyzed using a logistic regression model. The model included binary status of whether or not a participant achieved their maximum possible reduction of OCS dose per protocol at Week 24 as the response variable, treatment groups, optimized OCS dose at baseline, regions, and baseline eosinophil level subgroups as covariates. Missing data was imputed by using a pattern mixture model by multiple imputation approach; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0024, Regression, Logistic — Threshold for significance at 0.05; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.4 to 4.73] — Dupilumab 300 mg q2w v Placebo q2w

6. Secondary Outcome: Percentage of Participants Who No Longer Required Oral Corticosteroids Dose at Week 24 While Maintaining Asthma Control
Description: Participants were classified according to the binary status of whether or not the participant still required OCS at Week 24 while maintaining asthma control.
Time Frame: Week 24
Population: Analysis was performed on ITT population with baseline OCS dose less than or equal to 30 mg/day.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 106 | 103
percentage of participants | 29.2 | 52.4
Statistical Analysis 1: Comparison: Placebo q2w vs Dupilumab 300 mg q2w; The outcome measure was analyzed using a logistic regression model. The model included the binary status of whether or not a participant no longer required OCS at Week 24 as the response variable, and treatment groups, optimized OCS dose at baseline, regions, and baseline eosinophil level subgroups as covariates. Missing data was imputed using a pattern mixture model by multiple imputation approach; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0015, Regression, Logistic — Threshold for significance at 0.05; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.47 to 5.1] — Dupilumab 300 mg q2w v Placebo q2w

7. Secondary Outcome: Absolute Reduction From Baseline in Oral Corticosteroids Dose at Week 24 While Maintaining Asthma Control
Description: Absolute reduction was calculated by subtracting Week 24 value from baseline value.
Time Frame: Baseline and Week 24
Population: Analysis was performed on ITT population but not included in the hierarchical testing procedure. Here, "number analyzed"= participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
mg/day
  Baseline | 11.75 (6.31) | 10.75 (5.90)
  Week 24: number analyzed (Participants) | 106 | 101
  Week 24 | 6.32 (6.75) | 3.13 (5.44)
  Absolute reduction at Week 24: number analyzed (Participants) | 106 | 101
  Absolute reduction at Week 24 | 5.45 (6.80) | 7.66 (6.10)

8. Other Pre Specified Outcome: Annualized Rate of Severe Exacerbation Events During The 24-Week Treatment Period
Description: A severe asthma exacerbation event was defined as a deterioration of asthma during the 24-week treatment period requiring: use of systemic corticosteroids for >=3 days (at least double the dose currently used); and/or hospitalization related to asthma symptoms or emergency room visit because of asthma requiring intervention with a systemic corticosteroid treatment. Annualized event rate was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 24
Population: Analysis was performed ITT population.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
Exacerbation per participant-year | 1.597 [1.248 to 2.043] | 0.649 [0.442 to 0.955]

9. Other Pre Specified Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Weeks 12 and 24
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on ITT population. Here, "number analyzed"= participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
liter
  Baseline | 1.63 (0.61) | 1.53 (0.53)
  Week 12: number analyzed (Participants) | 105 | 99
  Week 12 | 1.68 (0.61) | 1.82 (0.63)
  Change at Week 12: number analyzed (Participants) | 105 | 99
  Change at Week 12 | 0.06 (0.50) | 0.29 (0.43)
  Week 24: number analyzed (Participants) | 104 | 97
  Week 24 | 1.63 (0.65) | 1.84 (0.60)
  Change at Week 24: number analyzed (Participants) | 104 | 97
  Change at Week 24 | 0.00 (0.51) | 0.29 (0.46)

10. Other Pre Specified Outcome: Change From Baseline in Asthma Control Questionnaire 5-Question Version (ACQ-5) Score at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: The ACQ-5 has 5 questions, reflecting top-scoring 5 asthma symptoms: woken at night by symptoms, wake in mornings with symptoms, limitation of daily activities, shortness of breath and wheeze. Participants were asked to recall how their asthma had been during previous week and to respond to each of 5 symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). ACQ-5 total score was mean of scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated lower asthma control.
Time Frame: Baseline and at Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Analysis was performed on ITT population. Here, number analyzed = participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
score on a scale
  Change at Week 2: number analyzed (Participants) | 102 | 95
  Change at Week 2 | -0.18 (0.67) | -0.49 (0.86)
  Change at Week 4: number analyzed (Participants) | 103 | 93
  Change at Week 4 | -0.36 (0.81) | -0.61 (1.01)
  Change at Week 8: number analyzed (Participants) | 104 | 96
  Change at Week 8 | -0.39 (1.13) | -0.68 (1.06)
  Change at Week 12: number analyzed (Participants) | 101 | 96
  Change at Week 12 | -0.54 (1.17) | -0.92 (1.09)
  Change at Week 16: number analyzed (Participants) | 104 | 95
  Change at Week 16 | -0.57 (1.05) | -0.87 (1.18)
  Change at Week 20: number analyzed (Participants) | 102 | 97
  Change at Week 20 | -0.53 (1.09) | -0.83 (1.19)
  Change at Week 24: number analyzed (Participants) | 99 | 96
  Change at Week 24 | -0.57 (1.19) | -0.94 (1.22)

11. Other Pre Specified Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Global Score at Week 12 and Week 24
Description: AQLQ is a disease-specific, self-administered quality of life questionnaire designed to measure functional impairments that were most important to participants with asthma. AQLQ comprised of 32 items in 4 domains: symptoms (12 items), activity limitation (11 items), emotional function (5 items), environmental stimuli (4 items). Each item was scored on a 7-point likert scale (1=maximal impairment, 7=no impairment). The 32 items of the questionnaire were averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired at all). Higher scores indicate better quality of life.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
score on a scale
  Change at Week 12: number analyzed (Participants) | 105 | 98
  Change at Week 12 | 0.56 (1.08) | 0.78 (1.09)
  Change at Week 24: number analyzed (Participants) | 100 | 98
  Change at Week 24 | 0.56 (0.97) | 0.94 (1.17)

12. Other Pre Specified Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Scores at Week 12 and Week 24
Description: EQ-5D-5L is a standardized health-related quality of life questionnaire developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state. EQ-5D-5L-VAS records participant's self-rated health on a vertical VAS that allows them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable).
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 10
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
score on a scale
  Single Index: Change at Week 12: number analyzed (Participants) | 105 | 98
  Single Index: Change at Week 12 | 0.04 (0.20) | 0.03 (0.17)
  Single Index: Change at Week 24: number analyzed (Participants) | 100 | 98
  Single Index: Change at Week 24 | 0.05 (0.18) | 0.05 (0.18)
  VAS Score: Change at Week 12: number analyzed (Participants) | 105 | 98
  VAS Score: Change at Week 12 | 5.99 (16.85) | 9.34 (18.20)
  VAS Score: Change at Week 24: number analyzed (Participants) | 100 | 98
  VAS Score: Change at Week 24 | 4.16 (16.74) | 11.06 (17.60)

13. Other Pre Specified Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Total Score at Week 12 and Week 24
Description: The HADS is a general scale to detect states of anxiety and depression already used and validated in asthma, which includes HADS-A and HADS-D subscales. The instrument is comprised of 14 items: 7 related to anxiety (HADS-A) and 7 to depression (HADS-D). Each item on the questionnaire is scored from 0-3. And, the total score is the sum of the scores of the 14 items ranging from 0 (no symptoms) to 42 (severe symptoms), with higher scores indicating higher anxiety/depression complains.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 107 | 103
score on a scale
  Change at Week 12: number analyzed (Participants) | 105 | 98
  Change at Week 12 | -0.75 (5.50) | -2.13 (5.32)
  Change at Week 24: number analyzed (Participants) | 100 | 98
  Change at Week 24 | -0.99 (5.36) | -2.53 (5.98)

14. Other Pre Specified Outcome: Change From Baseline in Sino Nasal Outcome Test-22 (SNOT-22) Global Score at Week 12 and Week 24
Description: The SNOT-22 is a validated measure of health related quality of life in sino nasal disease. It is a 22 item questionnaire with each item assigned a score ranging from 0-5. The total score may range from 0 (no disease) -110 (worst disease), lower scores represent better health related quality of life.
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on ITT population with bilateral nasal polyposis/chronic rhinosinusitis. Here, number analyzed = participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 41 | 31
score on a scale
  Change at Week 12: number analyzed (Participants) | 38 | 29
  Change at Week 12 | -3.79 (21.34) | -12.45 (17.10)
  Change at Week 24: number analyzed (Participants) | 37 | 27
  Change at Week 24 | -2.46 (19.11) | -14.56 (15.89)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 36) regardless of seriousness or relationship to investigational product.
Description: Reported AEs were treatment emergent AEs developed/worsened occurred during 'treatment-emergent period' (from first dose of study drug injection until 98 days after last dose of drug) or entry in the LTS12551 study (NCT02134028). Analysis was performed on safety population which included all participants who actually received at least 1 dose or part of a dose of the IMP and analyzed according to the treatment that participants actually received.
Groups:
- Placebo q2w: Participants who received Placebo (for Dupilumab) in combination with OCS and stable ICS (mean exposure of 24 weeks).
- Dupilumab 300mg q2w: Participants who received Dupilumab 300 mg q2w in combination with OCS and stable ICS (mean exposure of 24 weeks).
Arm/Group | Placebo q2w | Dupilumab 300mg q2w
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/103
Serious Adverse Events (participants affected / at risk) | 6/107 | 9/103
Other Adverse Events (participants affected / at risk) | 30/107 | 29/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo q2w (N=107) | Dupilumab 300mg q2w (N=103)
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo q2w (N=107) | Dupilumab 300mg q2w (N=103)
Bronchitis (Infections and infestations) | 6 | 7
Influenza (Infections and infestations) | 6 | 3
Sinusitis (Infections and infestations) | 4 | 7
Viral upper respiratory tract infection (Infections and infestations) | 19 | 9
Eosinophil count increased (Investigations) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT02528214/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT02528214/SAP_001.pdf